CLINICAL TRIAL: NCT01836406
Title: Effect of Ketorolac and Remote Ischemic Preconditioning on Renal Ischemia-reperfusion Injury in Patients Undergoing Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0485
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Renal Cell Carcinoma
Keywords: ketorolac; remote ischemic preconditioning; partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keromin Group (Experimental)
  Interventions: Drug: Ketorolac tromethamine and remote ischemic preconditioning
- Placebo Group (Placebo Comparator)

INTERVENTIONS:
Drug: Ketorolac tromethamine and remote ischemic preconditioning — Ketorolac tromethamine/ single / 1mg/kg/ intravenous administration 30 min before renal artery clamping, remote ischemic preconditioning / 200 mmHg / 5 min inflation and 10 min deflation / 3 cycles / after anesthetic induction
  Arms: Keromin Group

SUMMARY:
Partial nephrectomy is a widely accepted alternative to radical nephrectomy in patients with clinically localized, unilateral renal cell carcinoma and a normal contralateral kidney. Interruption of renal blood flow via pedicle clamping is often necessary during partial nephrectomy, especially for complex tumors with deep parenchymal invasion. Ischemia-reperfusion injury is a complex process involving several mechanisms including renal vasoconstriction, extensive tubular damage and glomerular injury. The investigators will examine the postoperative renal function of patients who received intraoperative ketorolac and remote ischemic preconditioning during partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA l and ll
* age 20-65
* patients undergoing partial nephrectomy

Exclusion Criteria:

* preoperative liver or renal dysfunction,
* coagulopathy,
* chronic alcoholism,
* hypersensitivity of NSAID,
* history of warfarin,
* history of gastric ulcer

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
serum creatinine | at baseline, 2 hr, 12hr, 24 hr, 48 hr, 72 hr after clamping release

SECONDARY OUTCOMES:
Creatinine clearance | at baseline, 2 hr, 12hr, 24 hr, 48 hr, 72 hr after clamping release
urinary NAG | at base line, 2 hr, 12 hr after clamping release
serum NGAL | at base line, 2 hr, 12 hr after clamping release

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea